CLINICAL TRIAL: NCT05163782
Title: Validation of an Ankle Foot Orthosis With Anterior Support for Foot Drop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TOPMED (Other)
Collaborators: Turbomed Orthotics Inc. (Unknown); Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD-19-0276_OptOrPi
Record Dates: First submitted 2021-12-15; First posted 2021-12-20 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-03

CONDITIONS: Foot Drop
MeSH Terms: conditions — Peroneal Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- People with foot drop (Experimental): People with left or right foot drop
  Interventions: Device: New ankle foot orthosis with anterior support; Device: Ankle foot orthosis with anterior support; Device: Ankle foot orthosis from competitor 1; Device: Ankle foot orthosis from competitor 2

INTERVENTIONS:
Device: New ankle foot orthosis with anterior support — New ankle foot orthosis with anterior support developed by Turbomed
Device: Ankle foot orthosis with anterior support — Ankle foot orthosis with anterior support from Turbomed
Device: Ankle foot orthosis from competitor 1 — Ankle foot orthosis with posterior support from competitor 1
Device: Ankle foot orthosis from competitor 2 — Ankle foot orthosis with posterior support from competitor 2

SUMMARY:
The objective of this research is to compare the new ankle foot orthosis (AFO) with prior support developed by Turbomed, with the AFO with posterior support from Turbomed as well as two competing AFOs currently on the market.

With this research, we seek to answer the following questions:

* Is the new AFO as biomechanically efficient as the AFOs currently on the market?
* Is the new AFO more comfortable than the AFO currently on the market?
* Is the new AFO easier to put on and attach than the AFOs currently on the market?

ELIGIBILITY:
Inclusion Criteria:

* Foot drop following surgery or an accident (functional calf, without contracture and not spastic)
* Foot drop following a Cerebral Vascular Accident (with or without spasticity, mild to moderate)
* Ability to stand and walk alone without technical assistance
* Ability to communicate comfort/discomfort

Exclusion Criteria:

* Sore to one of the feet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Knee flexion angle during gait | At delivery
  Maximum, minimum and range of motion of the knee flexion angle during gait.
Hip flexion angle during gait | At delivery
  Maximum, minimum and range of motion of the hip flexion angle during gait.
Minimum foot clearance | At delivery
  Minimum foot clearance is defined as the minimum distance between the foot and the ground during swing.
Comfort of participants with orthosis | At delivery
  Comfort is measured with a Likert scale from 1 (not comfortable) to 5 (very comfortable).
Easy to put on orthosis | At delivery
  Easy to put on is measured with a Likert scale from 1 (very difficult) to 5 (very easy).

CONTACTS AND LOCATIONS:
Overall Officials: Edith Martin, PhD, Principal Investigator — TOPMED
Locations (1):
- TOPMED, Québec, Quebec, Canada